CLINICAL TRIAL: NCT00866008
Title: The Impact of the Heterogeneity of the Recruited Cohort of Follicles During Ovarian Hyperstimulation for IVF on Aneuploidy Rates of Generated Embryos.
Brief Title: A Study of the Effects of a Novel Ovarian Stimulation Regimen on Embryo Aneuploidy Rates in In Vitro Fertilization (IVF)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to a very slow inclusion rate.
Sponsor: Bart CJM Fauser (Other)
Responsible Party: Sponsor-Investigator, Bart CJM Fauser, Professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOSTrial; CCMO: NL18499.000.07(a); METC: 07/172
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: In Vitro Fertilization
Keywords: IVF; In vitro implantation; Preimplantation genetic screening; Aneuploidy
MeSH Terms: conditions — Aneuploidy | interventions — Ovulation Induction; follitropin beta; ganirelix; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Conventional regimen with a daily dose of 225 IU recombinant FSH and GnRH agonist long protocol co-treatment.
  Interventions: Drug: Ovarian stimulation
- 2 (Experimental): Mild ovarian stimulation regimen using the endogenous FSH production by starting treatment on day 5 of the menstrual cycle with 150 IU / d recFSH with GnRH antagonist co treatment starting on day 6. As soon as two follicles reach 12 mm, treatment is continued with 200 IU / d rec hCG.
  Interventions: Drug: Ovarian stimulation

INTERVENTIONS:
Drug: Ovarian stimulation — 1. Conventional regimen with a daily dose of 225 IU recombinant FSH and GnRH agonist long protocol co-treatment
  2. Mild ovarian stimulation regimen using the endogenous FSH production by starting treatment on day 5 of the menstrual cycle with 150 IU / d recFSH with GnRH antagonist co treatment starting on day 6. As soon as two follicles reach 12 mm, treatment is continued with 200 IU / d rec hCG.
  Other Names: Follitropine (Puregon); Ganirelix (Orgalutran); Triptoreline (Decapeptyl)

SUMMARY:
Background:

By limiting the number of embryos transferred to the uterus to only a single embryo, the risk of multiple gestation can be reduced. In order to improve the effectiveness of single embryo transfer, the ability to select the embryo with the highest potential to develop into a healthy child is of vital importance. While embryos rated as high quality by standardized morphological assessment are associated with higher implantation and pregnancy rates, it is still not possible to predict with certainty which embryo will implant and has the highest potential to develop into a healthy child. An increasing body of evidence indicates that the incidence of chromosomal abnormalities in embryos is extremely high and good embryo morphology does not necessarily exclude an abnormal chromosomal constitution. Since aneuploidies are considered the main cause of embryonic wastage and loss, this phenomenon may be primarily responsible for the relatively poor pregnancy rates reported after IVF.

The introduction of fluorescent in-situ hybridization (FISH) techniques for preimplantation genetic diagnosis has enabled screening of embryos for chromosomal aneuploidies before transfer. Preimplantation genetic screening (PGS) would be of special interest for couples that are thought to have a higher risk of developing chromosomally abnormal embryos, with the aim of improving their chances for an ongoing pregnancy after IVF. PGS is applied clinically in numerous IVF laboratories throughout the world, and high rates of chromosomal abnormalities have been reported in IVF derived embryos. However, a recent meta-analysis has shown that PGS is yet to have a significant impact on IVF outcomes. This may partly be explained by the fact that most aneuploidies observed at this stage originate during the first mitotic divisions of early preimplantation development, resulting in chromosomally mosaic embryos. If a chromosomally mosaic embryo is biopsied, this cell may not be representative for the remaining embryo.

The investigators' group recently completed the first prospectively designed, randomized trial, comparing embryo aneuploidy rates following two ovarian hyperstimulation regimes in a group of 111 IVF patients. Milder stimulation was associated with a reduction in the number of oocytes retrieved and embryos generated. However, the proportion of chromosomally normal embryos was significantly increased. These results showed for the first time a direct correlation between the ovarian stimulation protocol and the incidence of chromosome abnormalities in the embryo. The observation that mild stimulation in some patients still resulted in a high oocyte yield and concurring higher proportions of abnormal embryos, underscores the need for further development of minimal stimulation approaches.

Primary Objective:

To determine whether the administration of hCG during the late follicular phase, instead of continuing with a fixed dose FSH, results in a more homogeneous cohort of growing follicles and the development of only the most competent oocytes, leading to lower aneuploidy rates in resulting embryos.

Study design:

Prospectively randomized, clinical study in 110 women undergoing IVF treatment

Intervention:

Randomization to one of two ovarian stimulation protocols:

1. Conventional regimen with a daily dose of 225 IU recombinant FSH and GnRH agonist long protocol co-treatment
2. Mild ovarian stimulation regimen using the endogenous FSH production by starting treatment on day 5 of the menstrual cycle with 150 IU / d recFSH with GnRH antagonist co treatment starting on day 6. As soon as two follicles reach 12 mm, treatment is continued with 200 IU / d rec hCG.

In both arms, oocyte pick up, insemination and embryo culture will be performed according to standard procedures. On day 3, all suitable embryos will be biopsied and one or two blastomeres removed, depending on the number of cells within the embryo.

FISH analysis will be performed for 10 chromosomes (1, 7, 13, 15, 16, 18, 21, 22, X and Y). Only chromosomally normal embryos will be transferred and cryopreserved. Embryos diagnosed as aneuploid or mosaic will be investigated for their implantation and developmental potential, by transferring them to an in vitro implantation model. After an extended culture period, implantation behaviour will be assessed and the entire embryo is reanalysed to detect the proportion of chromosomally abnormal cells. The implantation behaviour will be correlated to the type of abnormality and the chromosome(s) involved.

Primary outcome parameters:

Ovarian response, as assessed by the number of oocytes obtained and the proportion of chromosomally abnormal embryos per patient.

Secondary outcome parameters:

Number of oocytes retrieved, fertilization rates and proportion of morphologically high quality embryos on day 3.

Serum estradiol, LH, progesterone, androgen and hCG levels on cycle day 3 and day of hCG.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≤ 37 years
* BMI 18-29 kg/m2
* Regular cycle (25-35 days)
* Standard indication for IVF
* No major uterine abnormalities
* Written informed consent

Exclusion Criteria:

* Indication for IVF male factor with a total motile sperm count < 20x106
* ICSI or andrological indication
* Known abnormal (male or female) karyotype
* Oocyte donation
* One previous IVF treatment not resulting in embryo transfer
* History of recurrent abortion
* Medical contra indication for pregnancy or IVF treatment
* Relevant systemic disease
* Active substance abuse

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Proportion of chromosomally abnormal and mosaic day 3 embryos per patient based on PGS analysis. | 2 years

SECONDARY OUTCOMES:
Number of oocytes retrieved. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nick S Macklon, Prof, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Baart EB, Martini E, Eijkemans MJ, Van Opstal D, Beckers NG, Verhoeff A, Macklon NS, Fauser BC. Milder ovarian stimulation for in-vitro fertilization reduces aneuploidy in the human preimplantation embryo: a randomized controlled trial. Hum Reprod. 2007 Apr;22(4):980-8. doi: 10.1093/humrep/del484. Epub 2007 Jan 4. PMID 17204525